CLINICAL TRIAL: NCT04877639
Title: A Comparative Study on the Safety and Efficacy of Esmketamine Versus Dexmedetomidine During Drug Induced Sleep Endoscopy in Children With Positional Obstructive Sleep Apnea: A Consort-prospective, Randomized, Controlled Clinical Trial
Brief Title: Safety and Efficacy of Esmketamine Versus Dexmedetomidine
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhongnan Hospital (Other)
Responsible Party: Principal Investigator, Xuemin Song, associate professor, Zhongnan Hospital
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Other
Other Study IDs: XM Song
Record Dates: First submitted 2021-05-04; First posted 2021-05-07 (Actual); Last update posted 2022-08-22 (Actual); Status verified 2022-08

CONDITIONS: Osa Syndrome
Keywords: pediatrics ;Osa Syndrome
MeSH Terms: conditions — Carnevale syndrome | interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Esmketamine group (Active Comparator): Intravenous injection of 1.0mg/kg esmketamine was given, and nasal endoscopy was started 3 minutes later to maintain 1.0mg/kg/h esmketamine
  Interventions: Drug: Esmketamine,Dexmedetomidine
- Dexmedetomidine group (Active Comparator): Dexmedetomidine 1 μg/ kg at least 10 min after intravenous injection + maintain 1 μ After intravenous injection of dexmedetomidine 1 ug / kg, sufentanil 0.05 mg / kg was given 5 minutes
  Interventions: Drug: Esmketamine,Dexmedetomidine

INTERVENTIONS:
Drug: Esmketamine,Dexmedetomidine — Two different drugs were given to observe which of the two drugs was more suitable for DISE detection

SUMMARY:
A comparative study on the safety and efficacy of esmketamine versus Dexmedetomidine during drug induced sleep endoscopy in children with positional obstructive sleep apnea: A consort-prospective, randomized, controlled clinical trial

DETAILED DESCRIPTION:
Methods: Eighty ASA Ⅰ - Ⅱ patients aged 3-13 years underwent elective surgery under general anesthesia. No serious cardiovascular disease, no liver and kidney dysfunction, no central nervous system disease and mental disease. Patients undergoing tonsillectomy under general anesthesia were selected as the research objects.

80 patients were randomly divided into dexmedetomidine group D (n = 40) and ketamine Group K (n = 40). Both groups were given midazolam 0.2mg/kg intravenously

Group K: induction: intravenous injection of 1.0mg/kg esmketamine, nasal endoscopy started 3 minutes later, maintained 1.0mg/kg/h esmketamine;

Group D: induction: Dexmedetomidine 1 μ G / kg at least 10 min after intravenous injection + maintain 1 μ After 5 minutes of intravenous injection of dexmedetomidine 1 ug / kg, sufentanil 0.05 mg / kg was given.

Propofol 0.5 mg · kg-1 was injected intravenously when the patient had body movement

Heart rate (HR), mean arterial pressure (map), electrocardiogram (ECG), respiratory rate (RR), pulse oxygen saturation (%, SpO2) and BIS were recorded before (T1), during (T2), after (T3), 1 min after tracheal intubation (T4), 1 min after extubation (T5) and 30 min after extubation (T6).

3.2 onset and maintenance time: the time from administration to endoscopic examination (min); Recovery time (min)

3.3 observation and treatment of adverse reactions during and after dis

3.4 observe the sedation score of the two groups during the dis phase and the awake score 30 minutes after waking up

Objective To observe the application of dexmedetomidine and esmketamine in drug-induced sleep nasal endoscopy, and to explore the best medication scheme, so as to better guide clinical medication.

ELIGIBILITY:
Inclusion Criteria:

* Eighty ASA Ⅰ - Ⅱ patients aged 3-13 years underwent elective surgery under general anesthesia. No serious cardiovascular disease, no liver and kidney dysfunction, no central nervous system disease and mental disease. Patients undergoing tonsillectomy under general anesthesia were selected as the research objects.

Exclusion Criteria:

* ASA grade III and above, abnormal heart, lung, liver and kidney function before operation; There were central nervous system diseases and mental diseases, preoperative allergy to anesthetics (dexmedetomidine, esmketamine), family history of malignant high fever, tracheostomy and other artificial airway.

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2023-05-01 (Estimated)

PRIMARY OUTCOMES:
Onset time, Vital signs | 1 year
  Time from administration to operation;Heart rate, blood pressure and body movement during operation

CONTACTS AND LOCATIONS:
Overall Officials: Yuanzhen Zhang, professor, Study Chair — Wuhan University
Locations (1):
- Zhongnan Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yongping Z, Xinyi L, Aming S, Qiang X, Tianqi Z, Mengmeng S, Xiong C, Xuemin S. The safety and efficacy of esketamine in comparison to dexmedetomidine during drug-induced sleep endoscopy in children with obstructive sleep apnea hypopnea syndrome: A randomized, controlled and prospective clinical trial. Front Pharmacol. 2022 Dec 1;13:1036509. doi: 10.3389/fphar.2022.1036509. eCollection 2022. PMID 36532775